CLINICAL TRIAL: NCT05130736
Title: The Use of a Rehabilitation Robot in Patients With Post-COVID-19 Fatigue Syndrome
Brief Title: Rehabilitation Robot in Patients With Post-Coronavirus Disease (COVID-19) Fatigue Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: EGZOTech sp. z o.o. (Unknown); Szpital Wojewódzki w Poznaniu (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 514/21
Record Dates: First submitted 2021-09-03; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Post-Viral Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot (Experimental): Patients treated using a rehabilitation robot
  Interventions: Device: Robot rehabilitation
- Control (Active Comparator): Patients receiving traditional rehabilitation treatment (robot used only as assessment tool)
  Interventions: Device: Robot rehabilitation

INTERVENTIONS:
Device: Robot rehabilitation — Effectiveness of using a rehabilitation robot in post-COVID-19 rehabilitation

SUMMARY:
The aim of the study is to compare the effectiveness of two models of rehabilitation:

* traditional neurological rehabilitation, and
* neurological rehabilitation combined with a rehabilitation robot (Luna by EGZOTech).

An additional goal is to test the qualitative diagnostic reference using the surface electromyogram of the Luna robot (certified as a Medical Device) for functional diagnostics based on standardized clinical tests.

ELIGIBILITY:
Inclusion Criteria:

- patients discharged from Intensive Care Units after undergone ventilator therapy due to COVID-19

Exclusion Criteria:

* active medical condition (infections; tumors; rheumatological, metabolic, endocrine, autoimmunological, cardiovascular diseases)
* bipolar disorder
* dementia
* nutritional disorders
* addiction to alcohol or psychoactive substances
* severe obesity
* overtraining

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle fatigue assessment | Baseline, after 3 and after 8 weeks
  Raw robot measurement data (isometric contraction of the muscle for 60 s - biceps, quadriceps)
Change in isokinetic muscle force | Baseline, after 3 and after 8 weeks
  Raw robot measurement data (5 repetitions during measurement with LUNA)

SECONDARY OUTCOMES:
Change in functional physical ability 1 | Baseline, after 3 and after 8 weeks
  Functional Independence Measure
Change in functional physical ability 2 | Baseline, after 3 and after 8 weeks
  Barthel Index
Change in functional physical ability 3 | Baseline, after 3 and after 8 weeks
  Berg Balance Test
Change in functional physical ability 4 | Baseline, after 3 and after 8 weeks
  Short Physical Performance Battery
Change in cognitive ability 1 | Baseline, after 3 and after 8 weeks
  Addenbrooke's Cognitive Examination (ACE-III)
Change in cognitive ability 2 | Baseline, after 3 and after 8 weeks
  Montreal Cognitive Assessment
Change in the quality of life | Baseline, after 3 and after 8 weeks
  WHOQOL
Change in depressive symptoms | Baseline, after 3 and after 8 weeks
  Beck's Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Hojan, MD, PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zasadzka E, Tobis S, Trzmiel T, Marchewka R, Kozak D, Roksela A, Pieczynska A, Hojan K. Application of an EMG-Rehabilitation Robot in Patients with Post-Coronavirus Fatigue Syndrome (COVID-19)-A Feasibility Study. Int J Environ Res Public Health. 2022 Aug 20;19(16):10398. doi: 10.3390/ijerph191610398. PMID 36012033